CLINICAL TRIAL: NCT01687413
Title: Adjuvant De-escalation, Extracapsular Spread, P16+, Transoral (ADEPT) Trial for Oropharynx Malignancy
Brief Title: Post Operative Adjuvant Therapy De-intensification Trial for Human Papillomavirus-related, p16+ Oropharynx Cancer
Acronym: ADEPT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual and funding issues
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201207059
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Oropharyngeal Neoplasms
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Radiotherapy (Experimental): * Patients undergo postoperative IMRT once daily, 5 days a week, for 6 weeks. The prescribed radiotherapy dose will be 60 Gy in 2 Gy once-daily fraction size (total of 30 fractions).
  * Patients can consent to participate in either the randomized (physician chooses radiotherapy arm or radiotherapy & cisplatin arm) or non-randomized (patient chooses radiotherapy arm or radiotherapy & cisplatin arm) pathways
  Interventions: Radiation: Intensity-modulated radiation therapy (IMRT)
- Radiotherapy, cisplatin (Active Comparator): * Patients undergo postoperative IMRT once daily, 5 days a week, for 6 weeks. The prescribed radiotherapy dose will be 60 Gy in 2 Gy once-daily fraction size (total of 30 fractions)
  * Patients also receive cisplatin 40 mg/m2 IV on Days 1, 8, 15, 22, 29, and 36 of radiation therapy (6 doses for a total of 240 mg/m2).
  * Patients can consent to participate in either the randomized (physician chooses radiotherapy arm or radiotherapy & cisplatin arm) or non-randomized (patient chooses radiotherapy arm or radiotherapy & cisplatin arm) pathways
  Interventions: Radiation: Intensity-modulated radiation therapy (IMRT); Drug: Cisplatin

INTERVENTIONS:
Radiation: Intensity-modulated radiation therapy (IMRT)
Drug: Cisplatin
  Other Names: CACP, CDDP, CPDD, DDP, Neoplatin
  Arms: Radiotherapy, cisplatin

SUMMARY:
This clinical trial studies the intensity of adjuvant ("helper") therapy required in p16 positive oropharynx cancer patients, who have had all known disease removed surgically by a minimally invasive approach, and who have extracapsular spread in their lymph nodes. Patients can consent to participate in either the randomized (physician chooses radiotherapy arm or radiotherapy & cisplatin arm) or non-randomized (patient chooses radiotherapy arm or radiotherapy & cisplatin arm) pathways. After the surgery, receive either radiation alone, or radiation and weekly cis-platinum during therapy. Patients are then followed for cancer, functional and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically confirmed p16 positive squamous cell carcinoma of the oropharynx (OPSCC).
* Patient must have undergone transoral resection of their T1-4a oropharynx primary to a negative margin, and a neck dissection(s).
* Patient's disease must be pathological N-stage positive.
* Patient's disease must show extracapsular spread (ECS) in their nodal metastasis verified by central pathologist's review.
* Patients with synchronous primaries are included.
* Patients with unknown primaries are included if the diagnosis and resection of a primary site in the oropharynx is made from an endoscopic or robotic surgical procedure(s).
* Patients with recent excisional node biopsies/neck dissections are included if material is evaluable for extracapsular spread.
* Patient must be ≥ 21 years of age.
* ECOG performance status ≤ 2 (Karnofsky ≥60%).
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin <1.5 X upper normal institutional limit
  * AST(SGOT)/ALT(SGPT) ≤2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Patient (or legally authorized representative) must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Patient must not have pathologically N stage negative disease.
* Patient must not have outside nodal tissue from previous neck biopsy/neck dissections in which ECS cannot be confirmed or denied.
* Patient must not have a true unknown primary in which permanent section results are negative for malignancy in completely excised ipsilateral oropharyngeal tissue (palatine and lingual tonsil).
* Patient must not have distant metastatic disease at presentation.
* Patient must not have gross residual and/or microscopic disease present after surgery including re-resection(s), per the operative and pathology report.
* Patient must not have transoral robotic surgery (TORS) for a T3 or T4 primary tumor.
* Patient must not have a history of prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; noninvasive cancers (for example, carcinoma in situ of the oral cavity, larynx, breast or cervix are all permissible) are permitted even if diagnosed and treated < 3 years ago.
* Patient must not have had previous systemic chemotherapy for the study cancer. (Note: prior chemotherapy for a different cancer is allowable).
* Patient must not be receiving any other investigational agents.
* Patient must not have had any prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Patient must not have any life-threatening comorbid illnesses e.g. stroke with major sequelae or myocardial infarction/ unstable angina within the preceding 3 months or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient must not be pregnant or breastfeeding. If a woman of childbearing potential, patient must agree to use medically acceptable forms of contraception.

Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Rich, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiotherapy | Radiotherapy, Cisplatin
Started | 27 | 15
Completed | 26 | 11
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Not eligible | 0 | 2
Not completed — Patient withdrew before completing all radiotherapy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiotherapy | Radiotherapy, Cisplatin | Total
Number analyzed (Participants) | 27 | 15 | 42
Age, Continuous [Median (Full Range); unit: years] | 56 [41 to 74] | 55 [32 to 74] | 56 [32 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 24 | 12 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 15 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 26 | 14 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 15 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease-free Survival (DFS)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy | Radiotherapy, Cisplatin
Number analyzed (Participants) | 24 | 11
Participants | 24 | 10

2. Primary Outcome: Locoregional Control
Description: Rate of patients with no recurrence at original oropharyngeal site or in the neck nodal basins.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy | Radiotherapy, Cisplatin
Number analyzed (Participants) | 27 | 11
Participants | 26 | 9

3. Secondary Outcome: Rate of Distant Metastasis
Description: Assessed by biopsy or imaging-detected recurrent disease at sites away from the original primary and cervical zone.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy | Radiotherapy, Cisplatin
Number analyzed (Participants) | 27 | 11
Participants | 2 | 0

4. Secondary Outcome: Disease Specific Survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy | Radiotherapy, Cisplatin
Number analyzed (Participants) | 24 | 10
Participants | 24 | 10

5. Secondary Outcome: Number of Complications/Acute Toxicity by Organ Class
Description: -Assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Approximately 18 weeks
Population: One participant in each Arm did not have adverse events collected.
Measure: Number; unit: number of adverse events
Arm/Group | Radiotherapy | Radiotherapy, Cisplatin
Number analyzed (Participants) | 26 | 10
number of adverse events
  Blood and lymphatic system disorders | 5 | 12
  Cardiac disorders | 0 | 1
  Ear and labyrinth disorders | 11 | 4
  Eye disorders | 2 | 0
  Gastrointestinal disorders | 104 | 61
  General disorders | 38 | 17
  Immune system disorders | 1 | 0
  Infections and infestations | 7 | 2
  Injury, poisoning and procedureal complications | 31 | 9
  Investigations | 20 | 60
  Metabolism and nutrition disorders | 11 | 26
  Musculoskeletal and connective tissue disorders | 15 | 9
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 1 | 0
  Nervous system disorders | 48 | 29
  Psychiatric disorders | 16 | 9
  Respiratory, thoracic and mediastinal disorders | 34 | 14
  Skin and subcutaneous tissue disorders | 32 | 14
  Surgical and medical procedures | 3 | 0
  Vascular disorders | 11 | 6

6. Secondary Outcome: Change in Quality of Life as Measured by the MD Anderson Dysphagia Inventory
Description: * Each item is scored on a 5 point Likert scale (strongly disagree, disagree, no opinion, agree, strongly agree). Strongly agree = 1, Disagree = 2, No opinion = 3, Agree = 4, and Strongly Agree = 5
  * The lower the score the lower the quality of life
Time Frame: Baseline, 1 month, 6 months, 12 months, and 24 months
Population: Some participants were not analyzed as the participants did not complete the questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline - Radiotherapy; 1 Month - Radiotherapy; 6 Months - Radiotherapy; 12 Months - Radiotherapy; 24 Months - Radiotherapy: * Patients undergo postoperative IMRT once daily, 5 days a week, for 6 weeks. The prescribed radiotherapy dose will be 60 Gy in 2 Gy once-daily fraction size (total of 30 fractions).
  * Patients can consent to participate in either the randomized (physician chooses radiotherapy arm or radiotherapy & cisplatin arm) or non-randomized (patient chooses radiotherapy arm or radiotherapy & cisplatin arm) pathways
- Baseline - Radiotherapy + Cisplatin; 1 Month - Radiotherapy + Cisplatin; 6 Months - Radiotherapy + Cisplatin; 12 Months - Radiotherapy + Cisplatin; 24 Months - Radiotherapy + Cisplatin: * Patients undergo postoperative IMRT once daily, 5 days a week, for 6 weeks. The prescribed radiotherapy dose will be 60 Gy in 2 Gy once-daily fraction size (total of 30 fractions)
  * Patients also receive cisplatin 40 mg/m2 IV on Days 1, 8, 15, 22, 29, and 36 of radiation therapy (6 doses for a total of 240 mg/m2).
  * Patients can consent to participate in either the randomized (physician chooses radiotherapy arm or radiotherapy & cisplatin arm) or non-randomized (patient chooses radiotherapy arm or radiotherapy & cisplatin arm) pathways
Arm/Group | Baseline - Radiotherapy | Baseline - Radiotherapy + Cisplatin | 1 Month - Radiotherapy | 1 Month - Radiotherapy + Cisplatin | 6 Months - Radiotherapy | 6 Months - Radiotherapy + Cisplatin | 12 Months - Radiotherapy | 12 Months - Radiotherapy + Cisplatin | 24 Months - Radiotherapy | 24 Months - Radiotherapy + Cisplatin
Number analyzed (Participants) | 23 | 11 | 22 | 11 | 13 | 7 | 15 | 7 | 17 | 8
score on a scale
  My swallowing ability limits my day to day activities. | 3.2608696 (1.3888318) | 4.0000000 (1.0954451) | 4.1818182 (1.2203186) | 4.1818182 (1.1677484) | 4.3076923 (0.9473309) | 3.5714286 (1.5118579) | 4.5000000 (0.6504436) | 3.2857143 (1.6035675) | 3.9375000 (1.3889444) | 4.6250000 (0.5175492)
  I am embarrassed by my eating habits. | 3.5454545 (1.2993505) | 4.4545455 (0.8201995) | 4.1818182 (1.2587357) | 4.4545455 (0.5222330) | 4.3846154 (1.1208971) | 3.8571429 (0.6900656) | 4.4285714 (0.7559289) | 3.1428571 (1.2149858) | 4.1250000 (1.2041595) | 4.1250000 (0.6408699)
  Swallowing is more difficult at the end of the day. | 3.3636364 (1.4974726) | 4.5454545 (0.6875517) | 3.8095238 (1.3273676) | 4.0909091 (0.9438798) | 4.6153846 (0.8697185) | 3.8571429 (1.0690450) | 4.2857143 (1.1387288) | 4.1428571 (1.0690450) | 4.4000000 (0.9102590) | 4.7500000 (0.4629100)
  I do not feel self-conscious when I eat. | 3.3913043 (1.3395769) | 4.0909091 (1.2210279) | 3.9090909 (1.1087999) | 4.1818182 (0.9816498) | 4.3846154 (0.9607689) | 3.7142857 (1.1126973) | 4.0769231 (1.3204506) | 3.7142857 (1.2535663) | 3.6875000 (1.3022417) | 4.5000000 (0.7559289)
  I am upset by my swallowing problem. | 3.2272727 (1.6599431) | 2.0909091 (1.5135749) | 2.8636364 (1.6123173) | 2.6363636 (1.3618170) | 3.1538462 (1.6756170) | 2.2857143 (1.2535663) | 2.7857143 (1.6723347) | 3.1428571 (1.3451854) | 3.0625000 (1.7308476) | 3.2500000 (1.4880476)
  People have difficulty cooking for me. | 3.2173913 (1.5062452) | 3.9090909 (1.2210279) | 3.7727273 (1.3777766) | 4.2727273 (1.0090500) | 3.7692308 (1.4806444) | 3.1428571 (1.2149858) | 4.2142857 (1.1883131) | 3.7142857 (1.3801311) | 3.9375000 (1.3400871) | 4.1250000 (0.6408699)
  Swallowing takes great effort. | 3.0869565 (1.5049326) | 3.4545455 (1.2135598) | 3.9545455 (1.0455016) | 3.9090909 (1.2210279) | 3.6923077 (1.3155870) | 3.0000000 (1.1547005) | 3.9285714 (1.3847680) | 3.1428571 (1.5735916) | 3.5625000 (1.2632630) | 3.3750000 (1.4078860)
  I do not go out because of my swallowing problem. | 3.9130435 (0.9960396) | 4.6363636 (0.5045250) | 4.3181818 (0.9454837) | 4.1818182 (0.9816498) | 4.5384615 (0.8770580) | 3.8571429 (1.0690450) | 4.6428571 (0.6333237) | 4.1428571 (1.0690450) | 4.1875000 (1.0468206) | 4.2500000 (0.8864053)
  My swallowing difficulty has caused me to lose income. | 4.2608696 (1.0538842) | 3.9090909 (1.7002674) | 4.5000000 (0.7400129) | 4.3636364 (0.8090398) | 4.6153846 (0.6504436) | 4.0000000 (1.1547005) | 4.6428571 (0.6333237) | 3.8571429 (1.2149858) | 4.6000000 (0.6324555) | 4.5000000 (0.7559289)
  It takes me longer to eat because of my swallowing problem. | 2.5909091 (1.4690162) | 2.4000000 (1.4298407) | 3.1818182 (1.5625487) | 2.9090909 (1.7002674) | 3.0769231 (1.4978617) | 2.1428571 (0.8997354) | 3.5000000 (1.6052798) | 3.0000000 (1.9148542) | 2.8750000 (1.5438048) | 3.1250000 (1.6420806)
  People ask me, "Why can't you eat that?" | 4.0869565 (1.1246431) | 4.0000000 (1.1547005) | 4.0000000 (1.2344268) | 3.7272727 (1.3483997) | 4.1538462 (1.2810252) | 3.4285714 (1.1338934) | 4.2142857 (1.1883131) | 3.0000000 (1.6329932) | 4.1875000 (1.3275918) | 4.5000000 (0.9258201)
  Other people are irritated by my eating problem. | 4.2608696 (0.8643122) | 4.2727273 (1.0090500) | 4.5454545 (0.7385489) | 4.3636364 (0.8090398) | 4.6923077 (0.6304252) | 3.8571429 (0.6900656) | 4.5714286 (0.7559289) | 4.1428571 (0.8997354) | 4.3750000 (0.8062258) | 4.3750000 (0.9161254)

7. Secondary Outcome: Change in Cognitive Function as Measured by Cognitive Failures Questionnaire
Description: * 25 questions to assess the frequency in which participants experience cognitive failures including forgetfulness, distractibility, and false triggering
  * Answers range from 0 = never to 4 = very often
  * The higher the score the worse the cognitive failures the participant has experienced
Time Frame: Baseline, 1 month, 12 months, and 24 months
Population: Some participants were not analyzed as the participants did not complete the questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Radiotherapy | Baseline - Radiotherapy + Cisplatin | 1 Month - Radiotherapy | 1 Month - Radiotherapy + Cisplatin | 12 Months - Radiotherapy | 12 Months - Radiotherapy + Cisplatin | 24 Months - Radiotherapy | 24 Months - Radiotherapy + Cisplatin
Number analyzed (Participants) | 24 | 11 | 22 | 11 | 16 | 7 | 17 | 8
score on a scale
  Do you read something and find you haven't been thinking about it and must read it again? | 1.4166667 (0.9743076) | 1.3636364 (1.2060454) | 1.5454545 (1.0107646) | 1.2727273 (0.7862454) | 1.4666667 (0.9154754) | 2.1666667 (1.1690452) | 1.5625000 (0.7274384) | 1.5714286 (1.1338934)
  Do you find you forget why you went from one part of the house to the other? | 1.2083333 (0.9770927) | 1.0909091 (0.9438798) | 1.2727273 (1.1621744) | 1.0000000 (1.0000000) | 1.333333 (1.3451854) | 1.5000000 (0.8366600) | 1.4375000 (0.8920949) | 1.4285714 (1.2724180)
  Do you fail to notice signposts on the road? | 0.6666667 (0.9168313) | 0.3636364 (0.6741999) | 0.7272727 (0.9847319) | 0.5454545 (0.6875517) | 0.6666667 (0.6172134) | 0.8333333 (0.7527727) | 0.6250000 (0.6191392) | 0.8571429 (1.0690450)
  Do you find you confuse right and left when giving directions? | 0.3333333 (0.8681147) | 0.2727273 (0.4670994) | 0.4545455 (0.9116846) | 0.2727273 (0.6466698) | 0.2666667 (0.5936168) | 0.3333333 (0.5163978) | 0.3750000 (0.6191392) | 0.5714286 (0.7867958)
  Do you bump into people? | 0.2500000 (0.5316095) | 0.1818182 (0.4045199) | 0.3636364 (0.6579517) | 0.1818182 (0.6030227) | 0.4666667 (0.7432234) | 0.8333333 (1.3291601) | 0.3125000 (0.4787136) | 0.5714286 (0.9759001)
  Do you find you forget whether you've turned off a light or a fire or locked the door? | 0.9583333 (0.9990938) | 0.6363636 (0.6741999) | 0.8636364 (1.1252705) | 0.6363636 (0.6741999) | 1.1333333 (1.0600988) | 1.3333333 (0.5163978) | 0.7333333 (0.7037316) | 1.2857143 (0.9511897)
  Do you fail to listen to people's names when you are meeting them? | 1.7083333 (1.3014763) | 1.0909091 (1.3003496) | 1.8181818 (1.0970247) | 1.0909091 (1.0444659) | 2.0000000 (1.1952286) | 1.3333333 (1.0327959) | 1.6250000 (1.0246951) | 1.4285714 (1.2724180)
  Do you say something and realize afterwards that it might be taken as insulting? | 1.0000000 (1.0632191) | 0.9090909 (0.8312094) | 1.0000000 (1.1126973) | 0.8181818 (0.6030227) | 1.0666667 (0.7988086) | 1.0000000 (0.6324555) | 1.2500000 (1.0000000) | 0.8571429 (1.4638501)
  Do you fail to hear people speaking to you when you are doing something else? | 1.3750000 (1.3772215) | 1.2727273 (1.2720778) | 1.4090909 (1.0980108) | 1.0909091 (0.7006490) | 1.4000000 (0.9102590) | 1.8333333 (0.9831921) | 1.4375000 (1.0307764) | 1.5714286 (0.9759001)
  Do you lose your temper and regret it? | 0.9583333 (1.0417029) | 1.0000000 (0.7745967) | 1.0909091 (1.0649879) | 0.8181818 (0.6030227) | 0.8666667 (0.8338094) | 0.8333333 (0.7527727) | 0.8125000 (0.7500000) | 1.4285714 (1.2724180)
  Do you leave important letters unanswered for days? | 0.6666667 (1.0772203) | 0.6363636 (1.0269106) | 1.0000000 (1.0235326) | 0.4545455 (0.9341987) | 0.7857143 (0.9749613) | 0.8333333 (0.7527727) | 0.8125000 (0.7500000) | 1.0000000 (1.1547005)
  Do you find you forget which way to turn on a road you know well but rarely use? | 0.4782609 (0.9472239) | 0.4545455 (0.8201995) | 0.4090909 (0.9591212) | 0.5454545 (0.9341987) | 0.3333333 (0.6172134) | 0.5000000 (0.8366600) | 0.3125000 (0.4787136) | 0.2857143 (0.4879500)
  Do you fail to see what you want in a supermarket (although it's there)? | 0.6250000 (0.7696696) | 0.4545455 (0.5222330) | 0.9090909 (1.0649879) | 0.5454545 (0.6875517) | 1.0666667 (1.0997835) | 1.0000000 (0.6324555) | 0.8750000 (0.7187953) | 0.7142857 (0.4879500)
  Do you find yourself suddenly wondering whether you've used a word correctly? | 0.5833333 (0.7172815) | 0.6363636 (0.6741999) | 0.7727273 (1.0203556) | 0.6363636 (0.8090398) | 0.8000000 (0.8618916) | 0.6666667 (1.2110601) | 0.7500000 (0.6831301) | 0.8571429 (0.8997354)
  Do you have trouble making up your mind? | 0.9583333 (1.0826363) | 0.9090909 (1.0444659) | 1.0000000 (1.1126973) | 0.9090909 (0.9438798) | 0.9333333 (0.9611501) | 1.0000000 (1.0954451) | 1.0625000 (0.9287088) | 1.1428571 (1.2149858)
  Do you find you forget appointments? | 0.5833333 (0.9743076) | 0.5454545 (0.6875517) | 0.7727273 (1.1097755) | 0.6363636 (0.6741999) | 0.5333333 (0.8338094) | 0.8333333 (0.7527727) | 0.6250000 (0.6191392) | 1.0000000 (1.1547005)
  Do you forget where you put something like a newspaper or a book? | 1.0416667 (0.8064504) | 1.00000000 (0.8944272) | 1.1363636 (1.0371873) | 0.8181818 (0.7507572) | 1.4000000 (0.9102590) | 1.3333333 (0.5163978) | 1.1250000 (0.7187953) | 1.5714286 (1.3972763)
  Do you find you accidentally throw away the thing you want and keep what you meant to throw away? | 0.5416667 (1.0623668) | 0.1818182 (0.4045199) | 0.5454545 (1.0107646) | 0.1818182 (0.6030227) | 0.6666667 (0.7237469) | 0.3333333 (0.5163978) | 0.6250000 (0.7187953) | 0.5714286 (0.7867958)
  Do you daydream when you out to be listening to something? | 1.1250000 (1.0347232) | 1.2727273 (1.0090500) | 1.1818182 (1.0064726) | 0.9090909 (0.8312094) | 1.0000000 (0.9258201) | 0.8333333 (1.1690452) | 1.0000000 (0.7302967) | 0.8571429 (1.0690450)
  Do you find you forget people's names? | 1.8333333 (1.1671842) | 1.6363636 (1.5015144) | 1.8636364 (1.3556040) | 1.6363636 (1.1200649) | 2.0666667 (1.3345233) | 1.6666667 (1.0327956) | 1.8125000 (0.9105859) | 1.8571429 (1.3451854)
  Do you start doing one thing at home and get distracted into doing something else (unintentionally)? | 1.2500000 (1.1887151) | 1.0909091 (1.0444659) | 1.5454545 (1.1843131) | 1.0000000 (0.7745967) | 1.3333333 (1.1126973) | 2.3333333 (1.2110601) | 1.3125000 (0.9464847) | 1.4285714 (1.5118579)
  Do you find you can't quite remember something although it's on the tip of your tongue? | 1.4166667 (0.9743076) | 1.4545455 (1.2135598) | 1.8181818 (0.8528029) | 1.2727273 (0.9045340) | 1.7333333 (1.0327956) | 2.0000000 (0.6324555) | 1.6250000 (0.6191392) | 1.5714286 (1.3972763)
  Do you find you forget what you came to the shops to buy? | 0.8333333 (0.8164966) | 0.6363636 (0.8090398) | 1.1363636 (0.9902118) | 0.3636364 (0.6741999) | 1.2666667 (1.3345233) | 1.1666667 (0.9831921) | 0.7500000 (0.8563488) | 0.7142857 (0.4879500)
  Do you drop things? | 0.4583333 (0.7790276) | 0.8181818 (0.6030227) | 0.8181818 (1.0527227) | 0.6363636 (0.6741999) | 0.6666667 (0.6172134) | 1.3333333 (1.0327956) | 1.0000000 (0.8944272) | 0.8571429 (0.6900656)
  Do you find you can't think of anything to say? | 0.7916667 (0.9315329) | 0.5454545 (0.6875517) | 0.8636364 (1.1252705) | 0.9090909 (0.7006490) | 0.8000000 (0.8618916) | 1.1666667 (0.7527727) | 1.0000000 (0.9660918) | 1.0000000 (1.0000000)

8. Secondary Outcome: Change in Quality of Life as Measured by Neck Dissection Impairment Index (NDII)
Description: -The NDII consists of 10 questions; each with a 5 level ordinally scaled response option ranging from "not at all" to "a lot". The response for each item is then scored from 1 to 5, with 5 denoting higher quality of life (Not at all) and 1 being the least (A lot).
Time Frame: Baseline, 12 months, and 24 months
Population: Some participants were not analyzed as the participants did not complete the questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Radiotherapy | Baseline - Radiotherapy + Cisplatin | 12 Months - Radiotherapy | 12 Months - Radiotherapy + Cisplatin | 24 Months - Radiotherapy | 24 Months - Radiotherapy + Cisplatin
Number analyzed (Participants) | 23 | 11 | 16 | 7 | 17 | 8
score on a scale
  Neck or shoulder pain or discomfort | 1.6086957 (1.1175920) | 2.0909091 (1.2210279) | 1.4666667 (0.9904304) | 2.4285714 (1.5118579) | 1.3125000 (0.8732125) | 1.7500000 (1.2817399)
  Neck or shoulder stiffness | 1.4545455 (1.1433981) | 2.0000000 (1.2649111) | 1.0000000 (0.8451543) | 2.4285714 (1.5118579) | 1.1875000 (1.0468206) | 1.7500000 (1.3887301)
  Difficulty with self-care activities because of neck or shoulder | 0.8695652 (0.9197009) | 1.2727273 (1.1037127) | 0.3333333 (0.8164966) | 1.0000000 (1.0000000) | 0.2500000 (0.5773503) | 0.5000000 (1.4142136)
  Limited ability to life light objects because of your shoulder or neck | 0.6521739 (0.8846517) | 1.6363636 (1.4333686) | 0.4000000 (0.7367884) | 0.8571429 (1.0690450) | 0.2500000 (0.5773503) | 0.5000000 (0.7559289)
  Limited ability to lift heavy objects because of your shoulder or neck | 1.6086957 (1.3395769) | 2.2727273 (1.4206273) | 0.5333333 (0.9904304) | 1.5714286 (1.7182494) | 0.4666667 (0.8338094) | 0.8750000 (0.9910312)
  Limited ability to reach for objects because of your shoulder or neck | 1.2173913 (1.3802675) | 2.0909091 (1.5135749) | 0.5333333 (0.8338094) | 1.7142857 (1.6035675) | 0.5625000 (0.9639329) | 0.7500000 (1.0350983)
  Overall activity level because of your shoulder or neck | 1.0000000 (1.2431631) | 1.9090909 (1.5782614) | 0.5333333 (0.8338094) | 1.5714286 (1.5118579) | 0.3750000 (0.6191392) | 0.6250000 (0.7440238)
  Has the treatment of your neck affected your participation in social activities? | 0.7391304 (1.1368774) | 0.9090909 (1.2210279) | 0.0666667 (0.2581989) | 0.8571429 (0.8997354) | 0.1875000 (0.4031129) | 0.5000000 (1.0690450)
  Limited in ability to do leisure or recreational activities because of your neck or shoulder? | 1.0869565 (1.3788349) | 1.7272727 (1.4893562) | 0.2000000 (0.5606119) | 1.4285714 (1.2724180) | 0.2500000 (0.4472136) | 0.7500000 (1.1649647)
  Limited in ability to do work including work at home because of neck or shoulder discomfort or pain? | 1.1304348 (1.3916749) | 1.7272727 (1.6180797) | 0.2666667 (0.5936168) | 1.2857143 (1.1126973) | 0.1250000 (0.3415650) | 0.5000000 (1.0690450)

9. Secondary Outcome: Change in Quality of Life as Measured by University of Michigan Xerostomia Questionnaire
Description: * It contains 8 questions regarding dryness either during feeding or in the unstimulated state. Participants rate each item from 0 to 10, where 10 indicates the maximum dryness or discomfort due to dryness.
  * The higher the score the worse the participant's xerostomia
Time Frame: Baseline, 1 month, 6 months, 12 months, and 24 months
Population: Some participants were not analyzed as the participants did not complete the questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Radiotherapy | Baseline - Radiotherapy + Cisplatin | 1 Month - Radiotherapy | 1 Month - Radiotherapy + Cisplatin | 6 Months - Radiotherapy | 6 Months - Radiotherapy + Cisplatin | 12 Months - Radiotherapy | 12 Months - Radiotherapy + Cisplatin | 24 Months - Radiotherapy | 24 Months - Radiotherapy + Cisplatin
Number analyzed (Participants) | 24 | 11 | 21 | 11 | 14 | 7 | 17 | 7 | 17 | 8
score on a scale
  Rate your difficulty in talking due to dryness | 2.3333333 (2.4788964) | 1.3636364 (2.2033033) | 2.8095238 (2.9089353) | 3.9090909 (2.3855626) | 3.0000000 (2.9612887) | 4.8571429 (3.2366944) | 2.5625000 (2.8276905) | 3.5714286 (3.2071349) | 3.6875000 (2.9825884) | 3.1250000 (2.7998724)
  Rate your difficulty chewing due to dryness | 2.3913043 (2.2711457) | 1.4545455 (2.5831623) | 3.5238095 (2.6947922) | 3.1818182 (2.8219916) | 3.0714286 (2.4326082) | 4.5714286 (3.5523299) | 2.6250000 (2.2766935) | 3.7142857 (3.8606686) | 3.6250000 (2.9183329) | 2.7500000 (2.6592158)
  Rate your difficulty in swallowing solid food due to dryness | 2.6956522 (2.6532104) | 1.6363636 (2.8380531) | 3.4285714 (2.5994505) | 3.9000000 (2.9608557) | 3.5000000 (2.9807072) | 5.2857143 (3.5456210) | 3.3750000 (3.0304015) | 4.1428571 (3.5321651) | 4.1250000 (2.8722813) | 3.2500000 (3.0118812)
  Rate the frequency of your sleeping problems due to dryness | 1.7916667 (1.8876985) | 1.5454545 (2.8412545) | 3.2857143 (2.9179249) | 3.0000000 (2.8982753) | 1.7142857 (2.0542104) | 4.4285714 (2.8199966) | 2.2500000 (2.2656861) | 3.5714286 (3.1014590) | 2.6000000 (2.8485585) | 2.7500000 (2.4348658)
  Rate your mouth or throat dryness when eating food | 2.2173913 (2.1523037) | 1.8181818 (3.0271499) | 3.8571429 (2.9203718) | 3.7272727 (3.2277208) | 3.5000000 (2.8216198) | 5.7142857 (3.0394235) | 3.5000000 (3.0767949) | 4.0000000 (3.6968455) | 3.8750000 (3.0523215) | 3.3750000 (3.0207615)
  Rate your mouth or throat dryness while not eating | 2.1250000 (2.1931217) | 1.5454545 (2.3393861) | 3.8571429 (2.7979584) | 3.0909091 (2.1191765) | 2.6428571 (2.8177226) | 4.7142857 (2.4976179) | 3.2500000 (2.7446918) | 3.4285714 (3.4572216) | 3.7500000 (3.1517191) | 2.6250000 (2.7222627)
  Rate the frequency of sipping liquids to aid swallowing food | 3.1739130 (2.7741039) | 2.2727273 (3.1013194) | 5.1428571 (3.2293299) | 4.0000000 (3.4351128) | 5.0000000 (2.6602487) | 6.7142857 (2.6903708) | 5.0625000 (3.5864328) | 5.0000000 (3.6968455) | 5.3125000 (3.2397274) | 4.1250000 (3.6815175)
  Rate the frequency of sipping liquids for oral comfort when not eating | 2.9565217 (2.7216015) | 2.0909091 (2.8090762) | 4.6190476 (3.3388050) | 3.3636364 (2.9076701) | 3.4285714 (3.1553199) | 5.2857143 (2.7516229) | 3.8750000 (3.4229617) | 3.7142857 (3.7733401) | 4.0000000 (3.4448028) | 2.7500000 (3.3273756)

10. Secondary Outcome: Change in Hearing as Measured by Hearing Handicap Inventory - Adult
Description: * 11 item questionnaire to identify issues with hearing
  * Answers are yes = 4, sometimes = 2, and no = 0
  * The higher the score the more issues the participant has with hearing
Time Frame: Baseline, 1 month, and 12 months
Population: Some participants were not analyzed as the participants did not complete the questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Radiotherapy | Baseline - Radiotherapy + Cisplatin | 1 Month - Radiotherapy | 1 Month - Radiotherapy + Cisplatin | 12 Months - Radiotherapy | 12 Months - Radiotherapy + Cisplatin
Number analyzed (Participants) | 24 | 11 | 22 | 11 | 16 | 7
score on a scale
  Does a hearing problem cause you to feel embarrassed when you meet new people? | 0.2500000 (0.6079188) | 0.5454545 (0.9341987) | 0.2380952 (0.6248809) | 0.1818182 (0.6030227) | 0.1333333 (0.3518658) | 1.0000000 (1.0000000)
  Does a hearing problem cause you to feel frustrated when talking to members of your family? | 0.1250000 (0.4484272) | 0.1818182 (0.6030227) | 0.5238095 (0.8728716) | 0.3636364 (0.8090398) | 0.1333333 (0.3518658) | 0.7142857 (0.9511897)
  Do you have difficulty hearing or understanding co-workers or clients or customers? | 0.5000000 (0.8340577) | 1.0909091 (1.0444659) | 0.6666667 (0.9128709) | 1.0909091 (1.0444659) | 0.1333333 (0.3518658) | 1.7142857 (0.4879500)
  Do you feel that any difficulty with your hearing limits or hampers your personal or social life? | 0.1666667 (0.4815434) | 0.6363636 (0.9244163) | 0.3809524 (0.7400129) | 0.7272727 (1.0090500) | 0.2000000 (0.5606119) | 0.7142857 (0.9511897)
  Do you feel handicapped by a hearing problem? | 0.1250000 (0.4484272) | 0.5454545 (0.9341987) | 0.1428571 (0.4780914) | 0.3636364 (0.8090398) | 0.0666667 (0.2581989) | 0.7142857 (0.9511897)
  Does a hearing problem cause you difficulty in the movies or in the theater? | 0.1666667 (0.4815434) | 0.4545455 (0.8201995) | 0.5238095 (0.8728716) | 0.2727273 (0.6466698) | 0.1333333 (0.5163978) | 0.4285714 (0.7867958)
  Does a hearing problem cause you difficulty when in a restaurant with relatives or friends? | 0.2173913 (0.5997364) | 0.7272727 (0.9045340) | 0.6190476 (0.8646497) | 0.8181818 (0.9816498) | 0.2666667 (0.5936168) | 1.5714286 (0.7867958)
  Does a hearing problem cause you to attend religious services less often than you would like? | 0.0416667 (0.2041241) | 0.1818182 (0.6030227) | 0.0000000 (0.0000000) | 0.0000000 (0.0000000) | 0.0000000 (0.0000000) | 0.0000000 (0.0000000)
  Does a hearing problem cause you to have argments with family members? | 0.2500000 (0.6756639) | 0.1818182 (0.6030227) | 0.1000000 (0.4472136) | 0.1818182 (0.6030227) | 0.2666667 (0.7037316) | 0.1428571 (0.3779645)
  Does a hearing problem cause you difficulty when listening to TV or radio? | 0.3750000 (0.7109364) | 0.4545455 (0.8201995) | 0.8571429 (0.9636241) | 0.4545455 (0.8201995) | 0.4000000 (0.7367884) | 0.7142857 (0.9511897)
  Does a hearing problem cause you difficulty when visiting friends or relatives or neighbors? | 0.3333333 (0.7019641) | 0.6363636 (0.9244163) | 0.1904762 (0.5117663) | 0.4545455 (0.8201995) | 0.1333333 (0.3518658) | 0.7142857 (0.9511897)

11. Secondary Outcome: Change in Quality of Life as Measured by Scale of Subjective Total Taste Acuity
Description: * 1 question that asks about taste acuity
  * Answers are 0 = same taste acuity as before treatment; 1 = mild loss of taste acuity, but not inconvenient in daily life; moderate loss of taste acuity, and sometimes inconvenient in daily life; severe loss of taste acuity, and frequently inconvenient in daily life; and 4 = almost complete or complete loss of taste acuity
  * The higher the score the worse the participant's taste acuity
Time Frame: Baseline, 1 month, 6 months, and 12 months
Population: Some participants were not analyzed as the participants did not complete the questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Radiotherapy | Baseline - Radiotherapy + Cisplatin | 1 Month - Radiotherapy | 1 Month - Radiotherapy + Cisplatin | 6 Months - Radiotherapy | 6 Months - Radiotherapy + Cisplatin | 12 Months - Radiotherapy | 12 Months - Radiotherapy + Cisplatin
Number analyzed (Participants) | 24 | 11 | 22 | 11 | 14 | 7 | 16 | 7
score on a scale | 1.0833333 (1.1000659) | 0.9090909 (0.8312094) | 2.1363636 (1.0821255) | 2.9090909 (1.0444659) | 0.9285714 (0.7300459) | 2.4285714 (0.9759001) | 1.0000000 (0.7559289) | 1.5714286 (0.7867958)

12. Secondary Outcome: Change in Quality of Life as Measured by Speech Handicap Index
Description: * 31 questions regarding participant's speech and the effects of speech on his/her life
  * The answers for the first 30 questions range from 0 = never to 4 = always and the answers for the 31st question ranges from 0 = excellent to bad = 4
  * The higher the score the worse the participant's speech is affecting his/her life
Time Frame: Baseline and 12 months
Population: Some participants were not analyzed as the participants did not complete the questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Radiotherapy | Baseline - Radiotherapy + Cisplatin | 12 Months - Radiotherapy | 12 Months - Radiotherapy + Cisplatin
Number analyzed (Participants) | 24 | 11 | 16 | 7
score on a scale
  My speech makes it difficult for people to understand me | 1.9565217 (1.0215078) | 1.7272727 (0.9045340) | 1.3333333 (0.6172134) | 1.8333333 (1.3291601)
  I run out of air when I speak | 1.5000000 (0.7223151) | 1.4545455 (0.6875517) | 1.2666667 (0.7037316) | 1.8333333 (1.3291601)
  The intelligibility of my speech varies throughout the day | 2.0000000 (1.0632191) | 1.5454545 (0.8201995) | 1.4000000 (0.7367884) | 1.8333333 (1.3291601)
  My speech makes me feel incompetent | 1.3750000 (0.6468990) | 1.2727273 (0.6466698) | 1.1333333 (0.3518658) | 1.5000000 (0.8366600)
  People ask me why I'm hard to understand | 1.2916667 (0.6240935) | 1.1818182 (0.4045199) | 1.1333333 (0.3518658) | 1.3333333 (0.5163978)
  I feel annoyed when people ask me to repeat | 1.3750000 (0.8242256) | 1.2727273 (0.6466698) | 1.3333333 (0.4879500) | 1.6666667 (1.0327956)
  I avoid using the phone | 1.6250000 (1.2091139) | 1.5454545 (0.9341987) | 1.1333333 (0.3518658) | 1.6666667 (1.0327956)
  I'm tense when talking to others because of my speech | 1.4166667 (0.7172815) | 1.5454545 (0.8201995) | 1.0666667 (0.2581989) | 1.6666667 (1.0327956)
  My articulation is unclear | 1.8333333 (0.9630868) | 1.8181818 (1.3506205) | 1.4666667 (0.7432234) | 1.8333333 (1.3291601)
  People have difficulty understanding me in a noisy room | 1.8750000 (1.0347232) | 1.8181818 (0.9816498) | 1.6000000 (0.9856108) | 1.8333333 (0.9831921)
  I tend to avoid groups of people because of my speech | 1.2500000 (0.6079188) | 1.727277 (0.9045340) | 1.2666667 (0.7988086) | 1.8333333 (1.3291601)
  People seem irritated with my speech | 1.1250000 (0.3378320) | 1.3636364 (0.5045250) | 1.1333333 (0.3518658) | 1.5000000 (0.8366600)
  People ask me to repeat myself when speaking face-to-face | 1.5416667 (0.7790276) | 1.7272727 (0.9045340) | 1.3333333 (0.4879500) | 1.8333333 (0.9831921)
  I speak with friends and neighbors and relatives less often because of my speech | 1.4166667 (0.7172815) | 1.2727273 (0.6466698) | 1.2666667 (0.7988086) | 1.5000000 (0.8366600)
  I feel ask though I have to strain to speak | 1.833333 (0.9630868) | 1.9090909 (1.1361818) | 1.2000000 (0.5606119) | 2.0000000 (1.2649111)
  I find other people don't understand my speaking problem | 1.1666667 (0.3806935) | 1.2727273 (0.6466698) | 1.0666667 (0.2581989) | 1.3333333 (0.5163978)
  My speaking difficulties restrict my person and social life | 1.3750000 (0.6468990) | 1.2727273 (0.6466698) | 1.2000000 (0.5606119) | 1.5000000 (0.8366600)
  The intelligibility is unpredictable | 1.5833333 (0.8805466) | 1.3636364 (0.8090398) | 1.1333333 (0.3518658) | 1.5000000 (0.8366600)
  I feel left out of conversations because of my speech | 1.2083333 (0.4148511) | 1.3636364 (0.6741999) | 1.3333333 (0.8164966) | 1.4285714 (0.7867958)
  I use a great deal of effort to speak | 1.8750000 (0.9469631) | 1.6363636 (0.9244163) | 1.2666667 (0.4577377) | 1.8571429 (1.0690450)
  My speech is worse in the evening | 1.6250000 (0.8753881) | 1.6363636 (0.9244163) | 1.3333333 (0.7237469) | 1.8571429 (0.8997354)
  My speech problem causes me to lose income | 1.2916667 (0.6902531) | 1.8181818 (1.2504545) | 1.0000000 (0.0000000) | 1.4285714 (0.7867958)
  I try to change my speech to sound different | 1.2916667 (0.8064504) | 1.0909091 (0.3015113) | 1.0666667 (0.2581989) | 1.2857143 (0.7559289)
  My speech problem upsets me | 1.2083333 (0.4148511) | 1.5454545 (0.8201995) | 1.2666667 (0.4577377) | 1.8571429 (1.0690450)
  I am less outgoing because of my speech problem | 1.2500000 (0.5316095) | 1.4545455 (0.6875517) | 1.0666667 (0.2581989) | 1.4285714 (0.7867958)
  My family has difficulty understanding me when I call them throughout the house | 1.5000000 (0.7801895) | 1.6363636 (0.8090398) | 1.1333333 (0.5163978) | 1.5714286 (0.9759001)
  My speech makes me feel handicapped | 1.3333333 (0.7019641) | 1.4545455 (0.6875517) | 1.0666667 (0.2581989) | 1.5714286 (0.9759001)
  I have difficulties to continue a conversation because of my speech | 1.5000000 (0.7801895) | 1.5454545 (0.8201995) | 1.1333333 (0.3518658) | 1.8571429 (1.0690450)
  I feel embarrassed when people ask me to repeat | 1.2083333 (0.5089774) | 1.3636364 (0.9244163) | 1.0000000 (0.0000000) | 1.2857143 (0.4879500)
  I'm ashamed of my speech problem | 1.0833333 (0.2823299) | 1.2727273 (0.9045340) | 1.0000000 (0.0000000) | 1.2857143 (0.4879500)
  How do you rate your own speech at this moment? | 2.1304348 (0.9678631) | 1.4545455 (0.5222330) | 1.3846154 (0.6504436) | 1.5714286 (0.7867958)

13. Secondary Outcome: Change in Quality of Life as Measured by EORTC QLQ-C30
Description: * 30 questions designed to assess the quality of life of cancer patients
  * The first 28 questions have answers that range from 1=not at all to 4 = very much. The higher score indicates a worse quality of life
  * The last 2 questions have answers that range from 1 = very poor to 7 = excellent. The higher score indicates a better quality of life
Time Frame: Baseline, 1 month, 6 months, 12 months, and 24 months
Population: Some participants were not analyzed as the participants did not complete the questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Radiotherapy | Baseline - Radiotherapy + Cisplatin | 1 Month - Radiotherapy | 1 Month - Radiotherapy + Cisplatin | 6 Months - Radiotherapy | 6 Months - Radiotherapy + Cisplatin | 12 Months - Radiotherapy | 12 Months - Radiotherapy + Cisplatin | 24 Months - Radiotherapy | 24 Months - Radiotherapy + Cisplatin
Number analyzed (Participants) | 24 | 11 | 22 | 11 | 14 | 7 | 16 | 7 | 17 | 8
score on a scale
  Do you have trouble doing strenuous activities, like carrying a heavy shopping bag or a suitcase? | 2.0000000 (0.9534626) | 2.0000000 (0.6324555) | 1.7727273 (0.9223065) | 1.4545455 (0.6875517) | 1.3571429 (0.6333237) | 1.7142857 (0.7559289) | 1.2666667 (0.5936168) | 1.5714286 (0.7867958) | 1.4375000 (0.6291529) | 1.6250000 (0.5175492)
  Do you have any trouble taking a long walk? | 1.7500000 (0.9440892) | 1.0909091 (0.6015113) | 1.3636364 (0.5810872) | 1.2727273 (0.4670994) | 1.2142857 (0.4258153) | 1.1428571 (0.3779645) | 1.2666667 (0.4577377) | 1.1428571 (0.3779645) | 1.2500000 (0.4472136) | 1.2500000 (0.4629100)
  Do you have any trouble taking a short walk outside of the house? | 1.0833333 (0.2823299) | 1.0000000 (0.0000000) | 1.0454545 (0.2132007) | 1.0000000 (0.0000000) | 1.0714286 (0.2672612) | 1.1428571 (0.3779645) | 1.0000000 (0.0000000) | 1.1428571 (0.3779645) | 1.0000000 (0.0000000) | 1.1250000 (0.3535534)
  Do you need to stay in bed or a chair during the day? | 1.4583333 (0.8329709) | 1.0000000 (0.0000000) | 1.2272727 (0.5284135) | 1.0909091 (0.3015113) | 1.1428571 (0.3631365) | 1.2857143 (0.4879500) | 1.2666667 (0.4577377) | 1.2857143 (0.4879500) | 1.1875000 (0.5439056) | 1.0000000 (0.0000000)
  Do you need help with eating, dressing, washing yourself or using the toilet? | 1.0833333 (0.2823299) | 1.0909091 (0.3015113) | 1.0909091 (0.4264014) | 1.0000000 (0.0000000) | 1.0714286 (0.2672612) | 1.1428571 (0.3779645) | 1.0000000 (0.0000000) | 1.2857143 (0.4879500) | 1.0000000 (0.0000000) | 1.0000000 (0.0000000)
  Were you limited in doing either your work or other daily activities? | 2.0833333 (1.0179548) | 1.6363636 (1.0269106) | 1.4090909 (0.7341397) | 1.2727273 (0.6466698) | 1.4285714 (0.6462062) | 1.1428571 (0.3779645) | 1.2000000 (0.5606119) | 1.2857143 (0.4879500) | 1.3750000 (0.8062258) | 1.0000000 (0.0000000)
  Were you limited in pursuing your hobbies or other leisure time activities? | 2.0000000 (1.0215078) | 1.6363636 (1.0269106) | 1.4545455 (0.7385489) | 1.4545455 (0.6875517) | 1.2857143 (0.6112498) | 1.4285714 (0.7867958) | 1.1333333 (0.5163978) | 1.4285714 (0.7867958) | 1.2500000 (0.5773503) | 1.3750000 (0.7440238)
  Were you short of breath? | 1.2916667 (0.6240935) | 1.0000000 (0.0000000) | 1.1363636 (0.3512501) | 1.3636364 (0.5045250) | 1.1428571 (0.3631365) | 1.4285714 (0.7867958) | 1.2666667 (0.5936168) | 1.4285714 (0.7867958) | 1.1875000 (0.5439056) | 1.3750000 (0.5175492)
  Have you had pain? | 2.0000000 (0.7801895) | 1.7272727 (0.7862454) | 1.5000000 (0.5976143) | 1.7272727 (0.9045340) | 1.7142857 (0.8254203) | 1.8571429 (0.8997354) | 1.6000000 (0.7367884) | 1.8571429 (0.8997354) | 1.6875000 (0.7932003) | 2.0000000 (0.7559289)
  Did you need to rest? | 1.9166667 (0.8805466) | 1.5454545 (0.5222330) | 1.5909091 (0.7341397) | 1.6363636 (0.6741999) | 1.5000000 (0.7595545) | 1.7142857 (0.7559289) | 1.6000000 (0.7367884) | 1.8571429 (0.6900656) | 1.6875000 (0.7041543) | 1.6250000 (0.7440238)
  Have you had trouble sleeping? | 1.8333333 (0.8681147) | 2.2727273 (1.1908744) | 1.5454545 (0.6709817) | 1.6363636 (0.6741999) | 1.3571429 (0.6333237) | 2.4285714 (0.9759001) | 1.9333333 (0.9611501) | 2.0000000 (0.8164966) | 1.3750000 (0.6191392) | 2.1250000 (0.6408699)
  Have you felt weak? | 1.9166667 (0.9743076) | 1.8181818 (0.7507572) | 1.6818182 (0.8387271) | 1.4545455 (0.5222330) | 1.5384615 (0.8770580) | 1.4285714 (0.7867958) | 1.3333333 (0.6172134) | 1.5714286 (0.7867958) | 1.5625000 (0.7274384) | 1.3750000 (0.5175492)
  Have you lacked appetite? | 1.6956522 (0.8756703) | 1.6363636 (0.9244163) | 1.6363636 (0.7267314) | 1.3636364 (0.5045250) | 1.3571429 (0.6333237) | 1.2857143 (0.4879500) | 1.2000000 (0.5606119) | 1.2857143 (0.7559289) | 1.5000000 (0.8944272) | 1.1250000 (0.3535534)
  Have you felt nauseated? | 1.1666667 (0.6370221) | 1.3636364 (0.5045250) | 1.1818182 (0.5010811) | 1.1818182 (0.4045199) | 1.2142857 (0.4258153) | 1.1428571 (0.3779645) | 1.1333333 (0.5163978) | 1.0000000 (0.0000000) | 1.1875000 (0.4031129) | 1.0000000 (0.0000000)
  Have you vomited? | 1.0833333 (0.4082483) | 1.0000000 (0.0000000) | 1.0454545 (0.2132007) | 1.0000000 (0.0000000) | 1.0714286 (0.2672612) | 1.0000000 (0.0000000) | 1.0000000 (0.0000000) | 1.0000000 (0.0000000) | 1.0000000 (0.0000000) | 1.0000000 (0.0000000)
  Have you been constipated? | 1.5000000 (0.7801895) | 1.8181818 (1.0787198) | 1.6363636 (0.7895420) | 1.0909091 (0.3015113) | 1.2142857 (0.4258153) | 1.1428571 (0.3779645) | 1.1333333 (0.3518658) | 1.5714286 (0.9759001) | 1.4000000 (0.8280787) | 1.7500000 (1.1649647)
  Have you had diarrhea? | 1.0416667 (0.2041241) | 1.1818182 (0.4045199) | 1.1363636 (0.3512501) | 1.0000000 (0.0000000) | 1.1428571 (0.3631365) | 1.1428571 (0.3779645) | 1.2000000 (0.4140393) | 1.1428571 (0.3779645) | 1.0666667 (0.2581989) | 1.1250000 (0.3535534)
  Were you tired? | 2.0000000 (0.8846517) | 2.0000000 (0.7745967) | 1.181818 (0.7950061) | 1.7272727 (0.6466698) | 1.6428571 (0.8418974) | 1.8571429 (0.6900656) | 1.7333333 (0.8837151) | 2.1428571 (0.6900656) | 1.4375000 (0.6291529) | 1.7500000 (0.4629100)
  Did pain interfere with your daily activities? | 1.6666667 (0.8164966) | 1.7272727 (0.6466698) | 1.2380952 (0.6248809) | 1.3000000 (0.4830459) | 1.2857143 (0.6112498) | 1.4285714 (0.7867958) | 1.3333333 (0.6172134) | 1.5714286 (0.7867958) | 1.1333333 (0.3518658) | 1.0000000 (0.0000000)
  Have you had difficulty in concentrating on things, like reading a newspaper or watching television | 1.4583333 (0.7790276) | 1.2727273 (0.6466698) | 1.2857143 (0.5606119) | 1.2727273 (0.6466698) | 1.3571429 (0.7449463) | 1.5714286 (0.7867958) | 1.4000000 (0.9102590) | 1.5714286 (0.7867958) | 1.3125000 (0.6020797) | 1.2500000 (0.4629100)
  Did you feel tense? | 1.3750000 (0.6468990) | 1.5454545 (0.6875517) | 1.4090909 (0.5903262) | 1.2727273 (0.4670994) | 1.2857143 (0.4688072) | 1.5714286 (0.7867958) | 1.4000000 (0.8280787) | 1.4285714 (0.7867958) | 1.1875000 (0.4031129) | 1.7500000 (1.0350983)
  Did you worry? | 1.9166667 (0.7755316) | 2.0000000 (0.6324555) | 1.4545455 (0.5958006) | 1.2727273 (0.4670994) | 1.3571429 (0.4972452) | 2.0000000 (0.8164966) | 1.4000000 (0.8280787) | 2.0000000 (0.8164966) | 1.4375000 (0.7274384) | 2.0000000 (0.7559289)
  Did you feel irritable? | 1.4166667 (0.8297022) | 1.5454545 (0.5222330) | 1.4090909 (0.6661253) | 1.2727273 (0.6466698) | 1.1428571 (0.5345225) | 1.7142857 (0.9511897) | 1.3333333 (0.8164966) | 1.8571429 (0.6900656) | 1.3125000 (0.6020797) | 1.6250000 (0.9161254)
  Did you feel depressed? | 1.5416667 (0.8836272) | 1.4545455 (0.6875517) | 1.3181818 (0.5679004) | 1.1818182 (0.4045199) | 1.2142857 (0.4258153) | 1.5714286 (0.9759001) | 1.3333333 (0.8164966) | 1.7142857 (0.7559289) | 1.3125000 (0.6020797) | 1.5000000 (0.7559289)
  Have you had difficulty remembering things? | 1.4166667 (0.7172815) | 1.2727273 (0.4670994) | 1.5454545 (0.8004328) | 1.6363636 (0.5045250) | 1.7142857 (0.8254203) | 1.8571429 (0.8997354) | 1.6000000 (0.6324555) | 2.1428571 (0.8997354) | 1.4375000 (0.5123475) | 1.8750000 (0.6408699)
  Has your physical condition or medical treatment interfered with your family life? | 1.7916667 (0.8836272) | 1.5454545 (0.8201995) | 1.3181818 (0.7162311) | 1.3636364 (0.5045250) | 1.2142857 (0.4258153) | 1.4285714 (0.7867958) | 1.2000000 (0.4140393) | 1.5714286 (0.7867958) | 1.0625000 (0.2500000) | 1.1250000 (0.3535534)
  Has your physical condition or medical treatment interfered with your social activities? | 2.0416667 (0.9990938) | 1.9090909 (1.0444659) | 1.5909091 (0.7963662) | 1.7272727 (0.9045340) | 1.1428571 (0.3631365) | 1.7142857 (0.7559289) | 1.3333333 (0.6172134) | 1.5714286 (0.7867958) | 1.1250000 (0.3415650) | 1.3750000 (0.5175492)
  Has your physical condition or medical treatment caused you financial difficulties? | 1.5416667 (1.0206207) | 2.3636364 (1.2060454) | 1.5909091 (0.9591212) | 1.9090909 (1.0444659) | 1.7142857 (0.9944903) | 2.1428571 (1.0690450) | 1.4666667 (1.0600988) | 1.8571429 (0.8997354) | 1.4375000 (0.8139410) | 1.8750000 (0.9910312)
  How would you rate your overall health during the past week? | 5.2083333 (1.2846643) | 5.2727273 (0.7862454) | 5.4090909 (1.1815684) | 5.5454545 (0.8201995) | 5.9285714 (1.2688145) | 5.2857143 (1.1126973) | 6.0666667 (1.0327956) | 5.5714286 (1.1338934) | 5.7500000 (1.1832160) | 5.7500000 (0.7071068)
  How would you rate your overall quality of life during the past week? | 5.0416667 (1.3666578) | 5.1818182 (0.7507572) | 5.6363636 (1.2167660) | 5.6363636 (0.8090398) | 6.1428571 (1.3506205) | 5.4285714 (0.7867958) | 6.1333333 (1.0600988) | 5.7142857 (1.1126973) | 6.0000000 (1.0954451) | 6.0000000 (0.5345225)

ADVERSE EVENTS:
Time Frame: Adverse events were followed through 3 months following last date of study treatment (approximately 18 weeks)
Arm/Group | Radiotherapy | Radiotherapy, Cisplatin
All-Cause Mortality (participants affected / at risk) | 1/27 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/11
Other Adverse Events (participants affected / at risk) | 26/27 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy (N=27) | Radiotherapy, Cisplatin (N=11)
Xerostomia (Gastrointestinal disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy (N=27) | Radiotherapy, Cisplatin (N=11)
Anemia (Blood and lymphatic system disorders) | 2 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 7
Diarrhea (Gastrointestinal disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 11 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 5
Dysphagia (Gastrointestinal disorders) | 6 | 5
Mucositis oral (Gastrointestinal disorders) | 11 | 8
Nausea (Gastrointestinal disorders) | 5 | 9
Odynophagia (Gastrointestinal disorders) | 3 | 4
Oral pain (Gastrointestinal disorders) | 1 | 1
Salivary duct inflammation (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Chills (General disorders) | 1 | 1
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 6
Injection site reaction (General disorders) | 0 | 1
Localized edema (General disorders) | 2 | 1
Pain - oropharynx (General disorders) | 3 | 0
Pain-chest (non-cardiac) (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Hand infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Oral thrush (Infections and infestations) | 4 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 13 | 10
Alanine aminotransferase increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 9 | 10
Neutrophil count decreased (Investigations) | 0 | 6
Platelet count decreased (Investigations) | 0 | 9
Weight loss (Investigations) | 3 | 4
White blood cell decreased (Investigations) | 3 | 10
Anorexia (Metabolism and nutrition disorders) | 1 | 6
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 4
Hyponatremia (Metabolism and nutrition disorders) | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint range decrease (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 3 | 0
Anosmia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Dysarthria (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 13 | 7
Headache (Nervous system disorders) | 3 | 6
Paresthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dry nasal cavity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 9
Desquamation (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0
Hot flashes (Vascular disorders) | 1 | 0
Lymphedema (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT01687413/Prot_SAP_000.pdf